CLINICAL TRIAL: NCT00326495
Title: A Phase II Study of BAY 43-9006 (Sorafenib) in Combination With Cetuximab (Erbitux ) in EGFR Expressing Metastatic Colorectal Cancer (CRC)
Brief Title: BAY 43-9006 Plus Cetuximab to Treat Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alice Chen, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060164; 06-C-0164; NCT00343772 (obsolete NCT alias)
Record Dates: First submitted 2006-05-16; First posted 2006-05-17 (Estimated); Results first posted 2015-08-07 (Estimated); Last update posted 2017-07-24 (Actual); Status verified 2017-06

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Sorafenib; Cetuximab; Advanced Cancer; Phase II; Colorectal Cancer; Colon Cancer; Rectal Cancer; CRC; Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Cetuximab; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BAY 43-9006 & Cetuximab (Experimental): BAY 43-9006: Administered orally at a dose of 400 mg twice a day (BID). Cetuximab will be given intravenously (IV) at a dose of 400 mg/m^2 initially as a loading dose on week 2, followed by 250 mg/m^2 weekly starting on week 3
  Interventions: Drug: Cetuximab; Drug: BAY 43-9006

INTERVENTIONS:
Drug: Cetuximab — Cetuximab is a recombinant human/mouse chimeric monoclonal antibody which binds specifically to the extracellular domain of the epidermal growth factor receptor (epidermal growth factor receptor (EGFR), human epidermal growth factor receptor 1 (HER1), c-ErbB) in normal and tumor cells, and competitively inhibits the binding of epidermal growth factor (EGF) and other ligands, such as transforming growth factor-alpha.
  Other Names: Erbitux
Drug: BAY 43-9006 — Is a potent inhibitor of proto-oncogene c-Raf (c-raf), and wild-type and mutant proto-oncogene b-Raf (b-raf) in vitro
  Other Names: Sorafenib

SUMMARY:
Background:

* Colorectal cancer (CRC) is a major public health problem in the U.S. and worldwide, and 5-year survival with widespread metastatic disease is less than 5%.
* Expression of epidermal growth factor receptor (EGFR) or up-regulation of the gene occurs in the majority of CRC cases (60-80%).
* Therapies targeting EGFR, like cetuximab, have shown activity in the treatment of solid tumors like CRC.
* Cetuximab is FDA (Food and Drug Administration) approved for the treatment of EGFR-expressing CRC, but clinical responses to cetuximab are seen in only 10% of EGFR-expressing CRC.
* One possible mechanism of resistance to cetuximab could be KRAS (Kirsten rat sarcoma) mutations.
* Another major pathway implicated in colon carcinogenesis is the vascular endothelial growth factor (VEGF) pathway, which is involved in angiogenesis and is a validated target for therapy in CRC.
* BAY 43-9006 is both a Raf kinase inhibitor and an inhibitor of VEGF receptor (VEGFR2) tyrosine kinase.
* We hypothesize that the combined inhibition of EGFR, VEGFR2, and the Ras-(rapidly accelerated fibrosarcoma) Raf pathway will demonstrate promising clinical activity in CRC. Furthermore, in patients with mutant KRAS, combination of cetuximab with a drug that inhibits Raf kinase and acts downstream of Ras mutations, could restore tumor sensitivity to cetuximab.

Objectives:

* To determine the rate of response (complete response (CR) + partial response (PR) + stable disease (SD) for 4 months) and toxicity profile of combination of BAY 43-9006 and cetuximab in previously treated EGFR-expressing metastatic CRC in patients with mutant KRAS.
* To evaluate BAY 43-9006 pharmacokinetics & pharmacogenomics (CYP3A4/5 (cytochrome P450 3A4/5)).
* To evaluate for this combination treatment pharmacodynamics, effect on tumor vascularity and effect on angiogenic cytokines.

Eligibility:

* Adults with histologically or cytologically documented, measurable, EGFR-expressing metastatic CRC, which has recurred or progressed following at least one prior 5FU (Fluorouracil)-based combination chemotherapy regimen administered for the treatment of metastatic disease.
* Patients must be KRAS mutation-positive.

Design:

* BAY 43-9006 will be administered 400 mg by mouth twice daily
* Cetuximab will be administered as 400 mg/m^2 loading dose (week 1) followed by 250 mg/m^2 IV (intravenous) weekly.
* If procedure may be performed safely, tumor biopsy will be obtained prior to treatment and after 4 weeks of treatment.
* Optional positron emission tomography (PET)/computerized tomography (CT) imaging with 89Zr-labeled, EGFR-targeting antibody panitumumab may be performed to evaluate radiation dosimetry, safety, and tumor distribution prior to and following treatment with study agents.
* Patients will be evaluated for response every 8 weeks using the RECIST (Response Evaluation Criteria in Solid Tumors) criteria.
* This trial uses a phase II optimal design targeting a response rate as defined above of 20% in patients with mutant KRAS. Up to 49 patients may be treated.

DETAILED DESCRIPTION:
Background:

Colorectal cancer (CRC) is a major public health problem; 5-year survival with widespread metastatic disease is less than 5%. Expression of epidermal growth factor receptor (EGFR) or up-regulation of the gene occurs in 60-80% of cases. Therapies targeting EGFR, like cetuximab, have shown activity in the treatment of solid tumors like CRC.

Cetuximab is Food and Drug Administration (FDA) approved for the treatment of EGFR-expressing CRC, but clinical responses to cetuximab are seen in only 10% of EGFR-expressing CRC. Recent data strongly implicate KRAS (Kirsten rat sarcoma viral oncogene homolog) mutations as a mechanism of resistance to anti-EGFR antibody therapies such as cetuximab.

Another major pathway implicated in colon carcinogenesis is the vascular endothelial growth factor (VEGF) pathway, which is involved in angiogenesis and is a validated target for therapy in CRC. BAY 43-9006 is both a Raf kinase inhibitor and an inhibitor of VEGF receptor (VEGFR2) tyrosine kinase.

We hypothesize that the combined inhibition of EGFR, VEGFR2, and the Ras-Raf pathway will demonstrate promising clinical activity in CRC; furthermore, in patients with mutant KRAS, combination of cetuximab with a drug that inhibits Raf kinase and acts downstream of Ras mutations, could restore tumor sensitivity to cetuximab.

Objectives:

To determine the rate of response (CR (complete response) +PR (partial response) +SD (stable disease) for 4 months) and toxicity profile of combination of BAY 43-9006 and cetuximab in previously treated EGFR-expressing metastatic CRC in patients with mutant KRAS.

To evaluate BAY 43-9006 pharmacokinetics & pharmacogenomics (CYP3A4/5).

To evaluate for this combination treatment pharmacodynamics in tumor biopsies, effect on tumor vascularity, and effect on angiogenic cytokines.

Eligibility:

Adults with histologically or cytologically documented, measurable, EGFR-expressing metastatic CRC, which has recurred or progressed following at least one prior Fluorouracil (5FU)-based combination chemotherapy regimen administered for the treatment of metastatic disease.

Patients must be KRAS mutation-positive

Design:

BAY 43-9006 will be administered 400 mg by mouth twice daily. Cetuximab will be administered as 400 mg/m^2 loading dose (week 1) followed by 250 mg/m^2 intravenous (IV) weekly.

Optional PET (positron emission tomography) /CT (computed tomography) imaging with (89)Zr-labeled, EGFR-targeting antibody panitumumab may be performed to evaluate radiation dosimetry, safety, and tumor distribution prior to and following treatment with study agents.

Patients will be evaluated for response every 8 weeks using the Response Evaluation Criteria in Solid Tumor (RECIST) criteria.

This trial uses a phase II optimal design targeting a response rate as defined above of 20% in patients with mutant KRAS. Up to 49 patients may be treated.

Patients will be stratified by tumor KRAS status (wild type vs. codon 12/13 mutation in KRAS).

Optional correlative (89)Zr-panitumumab PET/CT imaging may be performed in up to 20 participants. For the first 5 patients, (89)Zr-panitumumab will be administered at baseline (within 10 days prior to starting cetuximab). PET/CT imaging will be performed up to 4 times: 2-6 hours following (89)Zr-panitumumab injection, 1-3 days following injection, 7-8 days following injection, and at the end of cycle 1/beginning of cycle 2, to obtain human dosimetry calculations.

If uptake into tumors is shown to be measurable in these first 5 patients, up to 15 subsequent

patients will be administered (89)Zr-panitumumab before cetuximab infusion (within 10 days prior to starting cetuximab) and have one PET/CT scan prior to the initial cetuximab infusion and a second (89)Zr-panitumumab infusion and scan at the end of cycle 1/beginning of cycle 2 (not shown in schema).

A diary will be provided for subjects to record taking study medication and side effects.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients must have histologically or cytologically documented metastatic colorectal cancer, which has recurred or progressed following at least one prior chemotherapy regimen administered for the treatment of metastatic disease. The diagnosis should be confirmed by the Laboratory of Pathology at the Clinical Center, NIH (National Institutes of Health).
* Tumor should express epidermal growth factor receptor (EGFR), defined as any membrane staining for EGFR in tumor cells by immunohistochemistry (IHC) done on archival tumor blocks or slides.
* Tumor blocks or unstained slides from archival pathological specimen suitable for the isolation of genomic DNA (deoxyribonucleic acid) must be available to determine the status of mutations in KRAS in the tumor. (For the initial 13 evaluable patients already enrolled and treated on this study, every effort will be made to re-acquire these blocks from patients or their referring physicians for evaluation of KRAS.)
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral computed tomography (CT) scan.
* Patients must have received or been offered and declined at least one prior Fluorouracil (5FU)-containing combination chemotherapy regimen for metastatic disease, unless available chemotherapy regimens were for some reason contraindicated for a particular patient. Patients who have received chemotherapy and/or biologic therapy, excluding BAY 43-9006 or cetuximab, are eligible. This therapy must have been completed greater than or equal to 4 weeks prior to enrollment on protocol, and the patient must have recovered to eligibility levels from prior toxicity. Prior radiation or surgery should have been completed greater than or equal to 4 weeks prior to study enrollment and all associated toxicities resolved to eligibility levels.
* Age greater than or equal to18 years. Colorectal cancer does not usually occur in patients less than 18 years of age.
* Life expectancy greater than 3 months.
* ECOG (Eastern Cooperative Oncology Group) performance status 0 or 1.
* Patients must have normal organ and marrow function as defined below:
* absolute neutrophil count greater than or equal to 1,500/ microliter
* platelets greater than or equal to 100,000/ microliter
* total bilirubin less than or equal to 1.5 times the institutional upper limits of normal
* AST (aspartate aminotransferase) (SGOT (serum glutamic oxaloacetic transaminase))/ALT (alanine aminotransferase) (SGPT (serum glutamic pyruvic transaminase) less than or equal to 2.5 times the institutional upper limit of normal
* creatinine less than or equal to 1.5 times the institutional upper limits of normal

OR

* creatinine clearance greater than or equal to 60 mL/min/1.73 m^2
* PT (prothrombin time)/PTT (partial thromboplastin time) less than or equal to 1.5 times the institutional upper limits of normal
* Patients must have at least one lesion amenable to biopsy, as determined by an associate investigator after discussion with a member of the interventional radiology team. This lesion should be different from target lesion(s) being followed on imaging studies to evaluate response to treatment.
* The effects of the combination of BAY 43-9006 and cetuximab on the developing human fetus at the recommended therapeutic doses are unknown. For this reason and because raf kinase inhibitor agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for at least 2 months following completion of study. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document and the ability to comply with daily oral self administration schedule.
* Patients must have systolic blood pressure less than or equal to 150 mm Hg and diastolic blood pressure less than or equal to 90 mmHg. Concomitant antihypertensive medications to achieve control of blood pressure are allowed.

EXCLUSION CRITERIA:

* Patients who have had chemotherapy, biologic therapy, or radiotherapy within 4 weeks prior to entering the study or those who have not recovered to at least eligibility levels from adverse events due to agents administered more than 4 weeks earlier. Patients must be greater than or equal to 2 weeks since any investigational agent administered as part of a Phase 0 study (also referred to as an early Phase I study or pre-Phase I study where a sub-therapeutic dose of drug is administered) at the PIs (principal investigator's) discretion, and should have recovered to eligibility levels from any toxicities
* Patients who have received any other investigational agents within 4 weeks prior to entering the study or those who have not recovered to at least eligibility levels from adverse events due to agents administered more than 4 weeks earlier.
* Patients with known brain metastases would be excluded from this clinical trial, with the exception of patients whose brain metastatic disease status remains stable for greater than or equal to 6 months after treatment of the brain metastases without steroids or anti seizure medications. These patients may be enrolled at the discretion of the principal investigator.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to BAY 43-9006 (for example, other multi-targeted kinase inhibitors, such as sunitinib) or cetuximab (for example, other drugs containing murine proteins, such as bevacizumab) used in the study.
* Prior therapy with cetuximab or BAY 43-9006.
* Patients on therapeutic anticoagulation are excluded. Prophylactic anticoagulation (i.e. low dose warfarin) of venous or arterial access devices is allowed provided that the requirements for PT, INR (International normalized ratio) or PTT are met.
* Evidence of bleeding diathesis.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active serious infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, uncontrolled hypertension, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because BAY 43-9006 is a kinase inhibitor agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with BAY 43-9006, breastfeeding should be discontinued if the mother is treated with BAY 43-9006.
* Human immunodeficiency virus (HIV)-positive patients receiving anti-retroviral therapy are excluded from this study due to the possibility of pharmacokinetic interactions between anti-retroviral medications and BAY 43-9006. HIV positive patients not receiving antiretroviral therapy are excluded due to the possibility that BAY 43-9006 may worsen their condition and the likelihood that the underlying condition may obscure the attribution of adverse events with respect to BAY 43-9006.
* History of another malignancy within the past 5 years, apart from adequately treated non-melanoma skin cancers, superficial bladder cancer or in situ cervical cancer.
* Patients with conditions that would impair their ability to swallow tablets are excluded.
* Use of the following medications will be not be allowed within 4 weeks prior to enrollment on the study and during the study: ketoconazole, itraconazole, ritonavir, cyclosporine, carbamazepine, phenytoin, phenobarbital, rifampin, St. Johns Wort, and prophylactic use of filgrastim and sargramostim. Products containing grapefruit juice will not be allowed while on study. BAY 43-9006 tosylate is metabolized by the P450 CYP3A enzyme; therefore, it is possible that BAY 43-9006 tosylate may interact with the above medications. Efforts should be made to switch patients who are taking enzyme-inducing anticonvulsant agents to other medications.
* Patients in whom resection is indicated and can be performed safely (unless surgery is declined by the patient for other reasons).
* For the optional PET/CT imaging with (89)Zr-panitumumab correlative study, participants with severe claustrophobia not relieved by oral anxiolytic medication or patients weighing > 136 kg (weight limit for scanner table).

Inclusion of Women and Minorities:

Both men and women and members of all races and ethnic groups are eligible for this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-05-10 (Actual); Primary Completion 2014-11-05 (Actual); Study Completion 2014-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shivaani Kummar, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cunningham D, Humblet Y, Siena S, Khayat D, Bleiberg H, Santoro A, Bets D, Mueser M, Harstrick A, Verslype C, Chau I, Van Cutsem E. Cetuximab monotherapy and cetuximab plus irinotecan in irinotecan-refractory metastatic colorectal cancer. N Engl J Med. 2004 Jul 22;351(4):337-45. doi: 10.1056/NEJMoa033025. PMID 15269313
- [Background] Messa C, Russo F, Caruso MG, Di Leo A. EGF, TGF-alpha, and EGF-R in human colorectal adenocarcinoma. Acta Oncol. 1998;37(3):285-9. doi: 10.1080/028418698429595. PMID 9677101
- [Background] Khosravi-Far R, Der CJ. The Ras signal transduction pathway. Cancer Metastasis Rev. 1994 Mar;13(1):67-89. doi: 10.1007/BF00690419. PMID 8143346
- [Result] Do K, Cao L, Kang Z, Turkbey B, Lindenberg ML, Larkins E, Holkova B, Steinberg SM, Raffeld M, Peer CJ, Figg WD, Eugeni M, Jacobs P, Choyke P, Wright JJ, Doroshow JH, Kummar S. A Phase II Study of Sorafenib Combined With Cetuximab in EGFR-Expressing, KRAS-Mutated Metastatic Colorectal Cancer. Clin Colorectal Cancer. 2015 Sep;14(3):154-61. doi: 10.1016/j.clcc.2015.02.007. Epub 2015 Mar 7. PMID 25861837
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2006-C-0164.html

RESULTS

PARTICIPANT FLOW:
Groups:
- BAY 43-9006 & Cetuximab: BAY 43-9006: Administered orally at a dose of 400 mg twice a day (BID)
  BAY 43-9006: is a potent inhibitor of proto-oncogene c-Raf (c-raf), and wild-type and mutant proto-oncogene b-Raf (b-raf) in vitro.
  Cetuximab will be given intravenously (IV) at a dose of 400 mg/m^2 initially as a loading dose on week 2, followed by 250 mg/m^2 weekly starting on week 3.
  Cetuximab is a recombinant human/mouse chimeric monoclonal antibody which binds specifically to the extracellular domain of the epidermal growth factor receptor (epidermal growth factor receptor (EGFR), human epidermal growth factor receptor 1 (HER1), c-ErbB) in normal and tumor cells, and competitively inhibits the binding of epidermal growth factor (EGF) and other ligands, such as transforming growth factor-alpha.
Period: Overall Study
Arm/Group | BAY 43-9006 & Cetuximab
Started | 51
Completed | 46
Not Completed | 5
Not completed — Switched to alternative treatment | 1
Not completed — Disease progression before treatment | 1
Not completed — Refused further treatment | 2
Not completed — Subject off study before assessment | 1

BASELINE CHARACTERISTICS:
Arm/Group | BAY 43-9006 & Cetuximab
Number analyzed (Participants) | 51
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 42
  >=65 years | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.65 (13.16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 46
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 36
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 51
Median Number of Previous Treatments [Median (Full Range); unit: Treatments] | 3 [1 to 5]

OUTCOME MEASURES:

1. Primary Outcome: Overall Rate of Response
Description: Rate of response is defined as the percentage of participants with a complete response (CR) + partial response (PR) + stable disease (SD) for 4 months. Response is defined by the Response is determined by the Response Evaluation Criteria in Solid Tumors (RECIST). Partial response is at least a 30% decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Complete response is a disappearance of all target lesions. Stable disease is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD (progressive disease), taking as reference the smallest sum LD since the treatment started. Progressive disease is at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 4 months
Population: Although 51 patients were accrued, only 50 were on study long enough for assessment.
Measure: Number; unit: percentage of participants
Arm/Group | BAY 43-9006 & Cetuximab
Number analyzed (Participants) | 50
percentage of participants | 15

2. Secondary Outcome: Count of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 96 months, 26 days
Population: Although 51 patients were accrued, only 50 were on study long enough for assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | BAY 43-9006 & Cetuximab
Number analyzed (Participants) | 50
Participants | 50

ADVERSE EVENTS:
Time Frame: 96 months, 26 days
Description: Although 51 patients were accrued, only 50 were on study long enough for assessment.
Arm/Group | BAY 43-9006 & Cetuximab
All-Cause Mortality (participants affected / at risk) | 2/50
Serious Adverse Events (participants affected / at risk) | 22/50
Other Adverse Events (participants affected / at risk) | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAY 43-9006 & Cetuximab (N=50)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Anaphylaxis (Immune system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bladder infection (Infections and infestations) | 2 (2)
Blood bilirubin increased (Investigations) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1)
Chills (General disorders) | 1 (1)
Death NOS (General disorders) | 2 (2)
Dehydration (Gastrointestinal disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Duodenal obstruction (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 5 (5)
Headache (Nervous system disorders) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (5)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Ischemia cerebrovascular (Nervous system disorders) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Movements involuntary (Nervous system disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 6 (6)
Tooth infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Wound infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BAY 43-9006 & Cetuximab (N=50)
Abdominal distension (Gastrointestinal disorders) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 14 (22)
Activated partial thromboplastin time prolonged (Investigations) | 17 (36)
Alanine aminotransferase increased (Investigations) | 33 (82)
Alkaline phosphatase increased (Investigations) | 31 (60)
Allergic reaction (Immune system disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Anal hemorrhage (Gastrointestinal disorders) | 1 (2)
Anal pain (Gastrointestinal disorders) | 1 (2)
Anemia (Blood and lymphatic system disorders) | 25 (62)
Anorexia (Metabolism and nutrition disorders) | 13 (19)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Ascites (Gastrointestinal disorders) | 6 (6)
Aspartate aminotransferase increased (Investigations) | 35 (92)
Ataxia (Nervous system disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6)
Bloating (Gastrointestinal disorders) | 2 (2)
Blood bilirubin increased (Investigations) | 21 (51)
Blurred vision (Eye disorders) | 2 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 5 (8)
Bruising (Injury, poisoning and procedural complications) | 1 (1)
Burn (Injury, poisoning and procedural complications) | 1 (1)
Buttock pain (Musculoskeletal and connective tissue disorders) | 1 (1)
CPK increased (Investigations) | 7 (13)
Catheter related infection (Infections and infestations) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 3 (3)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Chills (General disorders) | 9 (14)
Confusion (Psychiatric disorders) | 2 (2)
Conjunctivitis (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 10 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Creatinine increased (Investigations) | 6 (12)
Cystitis noninfective (Renal and urinary disorders) | 1 (1)
Cytokine release syndrome (Immune system disorders) | 7 (8)
Dehydration (Metabolism and nutrition disorders) | 10 (15)
Diarrhea (Gastrointestinal disorders) | 32 (152)
Dizziness (Nervous system disorders) | 4 (7)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 19 (19)
Dysgeusia (Nervous system disorders) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 5 (6)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 2 (3)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (7)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Extrapyramidal disorder (Nervous system disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fatigue (General disorders) | 25 (34)
Fever (General disorders) | 18 (36)
Flatulence (Gastrointestinal disorders) | 7 (10)
Flu like symptoms (General disorders) | 3 (4)
Flushing (Vascular disorders) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 22 (29)
Hematuria (Renal and urinary disorders) | 2 (2)
Hemoglobinuria (Renal and urinary disorders) | 3 (3)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (2)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 9 (14)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (6)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 5 (9)
Hypermagnesemia (Metabolism and nutrition disorders) | 8 (12)
Hypernatremia (Metabolism and nutrition disorders) | 4 (5)
Hypertension (Vascular disorders) | 16 (100)
Hyperuricemia (Metabolism and nutrition disorders) | 4 (8)
Hypoalbuminemia (Metabolism and nutrition disorders) | 42 (127)
Hypocalcemia (Metabolism and nutrition disorders) | 10 (14)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 17 (40)
Hypomagnesemia (Metabolism and nutrition disorders) | 26 (58)
Hyponatremia (Metabolism and nutrition disorders) | 30 (73)
Hypophosphatemia (Metabolism and nutrition disorders) | 34 (117)
Hypotension (Vascular disorders) | 1 (1)
Infections and infestations - Other,Upper airway NOS (Infections and infestations) | 1 (1)
Infusion related reaction (General disorders) | 3 (6)
Insomnia (Psychiatric disorders) | 3 (3)
Investigations - Other, specify (Investigations) | 6 (12)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1)
Lip infection (Infections and infestations) | 1 (2)
Lipase increased (Investigations) | 2 (3)
Lymphocyte count decreased (Investigations) | 33 (115)
Mucosal infection (Infections and infestations) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 13 (22)
Musculoskeletal and connective tissue disorder - Other, Restless leg (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 11 (12)
Nail loss (Skin and subcutaneous tissue disorders) | 1 (3)
Nausea (Gastrointestinal disorders) | 21 (51)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Neutrophil count decreased (Investigations) | 5 (17)
Non-cardiac chest pain (General disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (5)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 19 (30)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3)
Platelet count decreased (Investigations) | 21 (44)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Proteinuria (Renal and urinary disorders) | 5 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 19 (26)
Rash acneiform (Skin and subcutaneous tissue disorders) | 35 (68)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 20 (43)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 2 (2)
Scrotal pain (Reproductive system and breast disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Serum amylase increased (Investigations) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 4 (12)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (1)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 4 (5)
Syncope (Nervous system disorders) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 3 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 7 (9)
Urinary tract pain (Renal and urinary disorders) | 1 (1)
Urine discoloration (Renal and urinary disorders) | 2 (2)
Vaginal infection (Infections and infestations) | 1 (1)
Vascular disorders - Other, Ecchymosis (Vascular disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (3)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 9 (9)
Vomiting (Gastrointestinal disorders) | 20 (42)
Weight loss (Investigations) | 13 (13)
White blood cell decreased (Investigations) | 16 (49)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No